CLINICAL TRIAL: NCT00001533
Title: Treatment of T-Large Granular Lymphocyte (T-LGL) Lymphoproliferative Disorders With Cyclosporine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 960142; 96-H-0142
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2006-07-17 (Estimated); Status verified 1999-10

CONDITIONS: Anemia; Leukemia, T-Cell; Lymphocytosis; Neutropenia; Thrombocytopenia
Keywords: Anemia; Chronic T Cell Lymphocytosis with Neutropenia; Immunosuppression; Neutropenia; T-LGL Leukemia
MeSH Terms: conditions — Anemia; Leukemia, T-Cell; Lymphocytosis; Neutropenia; Thrombocytopenia; Leukemia, Large Granular Lymphocytic | interventions — Cyclosporine

INTERVENTIONS:
Drug: cyclosporine

SUMMARY:
T Cell Large Granular Lymphocyte (T-LGL) Lymphoproliferative Disorders are a heterogeneous group of uncommon diseases which may involve a polyclonal or a monoclonal T cell population, which bear characteristic surface markers corresponding to activated cytotoxic (CD3+, CD8+) lymphocytes. They are often associated with quite severe neutropenia, anemia, and thrombocytopenia which may be life-threatening. There is some evidence that the abnormal cytotoxic lymphocyte population may cause the cytopenias by suppressing hematopoiesis, although the mechanism is unclear. Case reports suggest that immunosuppressive therapy directed toward T cells may reverse the cytopenia. This pilot study involving up to 25 patients evaluates the clinical response to cyclosporine, an immunosuppressive drug, and seeks to elucidate the mechanism underlying the cytopenia.

DETAILED DESCRIPTION:
T Cell Large Granular Lymphocyte (T-LGL) Lymphoproliferative Disorders are a heterogeneous group of uncommon diseases which may involve a polyclonal or a monoclonal T cell population, which bear characteristic surface markers corresponding to activated cytotoxic (CD3+, CD8+) lymphocytes. They are often associated with quite severe neutropenia, anemia, and thrombocytopenia which may be life-threatening. There is some evidence that the abnormal cytotoxic lymphocyte population may cause the cytopenias by suppressing hematopoiesis, although the mechanism is unclear. Case reports suggest that immunosuppressive therapy directed toward T cells may reverse the cytopenia. This pilot study involving up to 25 patients evaluates the clinical response to cyclosporine, an immunosuppressive drug, and seeks to elucidate the mechanism underlying the cytopenia.

ELIGIBILITY:
Patients must be greater than or equal to 18 years of age.

Peripheral blood absolute LGL count of greater than or equal to 300/ul (performed on a manual differential), with LGL cells having the characteristic appearance of large lymphocytes with abundant pale blue cytoplasm, with or without a perinuclear clear zone, with varying degrees of azurophilic granules.

Immunophenotypic studies of peripheral blood showing an increased population of T-LGL (Staining for: CD3, CD8, and either CD16 or CD57+/- CD56).

Severe neutropenia (less than or equal to 500 neutrophils/uL of peripheral blood), or severe thrombocytopenia (less than or equal to 20,000 platelets/uL, or moderate thrombocytopenia (less than or equal to 50,000 platelets/uL with active bleeding , or anemia (hemoglobin less than or equal to 9 gm/dL), or red blood cell transfusion requirement of greater than or equal to 2 units/month for two months prior to initiation of CsA treatment.

Patients must not have had previous treatment with CsA or FK506.

Patients must not have a reactive LGL lymphocytosis to a viral infection.

Patients must not have a ECOG performance status of greater than 3.

Patients must not be currently pregnant, or unwilling to take oral contraceptives unless postmenopausal.

Mothers must not be breast feeding.

Patients must be able to give informed consent.

Patients must not be HIV positive.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1996-09; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Loughran TP Jr. Clonal diseases of large granular lymphocytes. Blood. 1993 Jul 1;82(1):1-14. PMID 8324214
- [Background] Witzig TE, Weitz JJ, Lundberg JH, Tefferi A. Treatment of refractory T-cell chronic lymphocytic leukemia with purine nucleoside analogues. Leuk Lymphoma. 1994 Jun;14(1-2):137-9. doi: 10.3109/10428199409049659. PMID 7920220
- [Background] Gabor EP, Mishalani S, Lee S. Rapid response to cyclosporine therapy and sustained remission in large granular lymphocyte leukemia. Blood. 1996 Feb 1;87(3):1199-200. No abstract available. PMID 8562948